CLINICAL TRIAL: NCT04279678
Title: Surgical Strategies in Moderate Ischemic Mitral Insufficiency in Patients Undergoing Coronary Artery Bypass Graft
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamad Zidane Roushdi, Principal Investigator, Assiut University
Other Study IDs: Moderate ischemic MR
Record Dates: First submitted 2020-02-18; First posted 2020-02-21 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Moderate Ischemic Mitral Regurgitation
MeSH Terms: interventions — Mitral Valve Annuloplasty; Coronary Artery Bypass

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- patients undergone mitral repair: includes all patients undergone repair of mitral valve with CABG
  Interventions: Procedure: Mitral valve repair
- patients with no mitral repair: includes all patients where no repair done for mitral valve , only CABG

INTERVENTIONS:
Procedure: Mitral valve repair — surgical repair of moderate ischemic mitral regurgitation using pericardial patch or rigid semi-annular ring
  Other Names: coronary artery bypass grafting
  Groups: patients undergone mitral repair

SUMMARY:
Ischemic mitral regurgitation (IMR) is a common complication of myocardial infarction, with a reported prevalence of 13-59%. Approximately one-third of these patients have at least moderate MR .

DETAILED DESCRIPTION:
Ischemic mitral regurgitation (IMR) is a common complication of myocardial infarction, with a reported prevalence of 13-59%. Approximately one-third of these patients have at least moderate MR .

The mechanism of IMR is complex and multifactorial.IMR results from the distortion and remodeling of the left ventricle after myocardial infarction ,where the papillary muscles are displaced away from the annular plane. Coupled with annular flattening, enlargement, and decreased contraction, this spatial deformation exerts traction on the chordae tendineae, leading to mal-coaptation of the structurally normal mitral valve and subsequently to secondary MR. Furthermore, the MR-related left ventricular(LV) volume overload promotes LV remodeling, resulting in exacerbation of the MR (MR begets more MR) . Two patterns of leaflet tethering have been reported in secondary MR: asymmetric tethering and symmetric tethering. Asymmetric tethering occurs with regional LV remodeling, resulting in displacement of the posterior papillary muscle in a lateral direction. Symmetric tethering generally results from global LV remodeling, resulting in apical tethering of both the anterior and posterior papillary muscles.

Most studies show that severe IMR is not usually improved by revascularization alone and that residual MR is associated with an increased mortality risk. It is generally accepted that severe IMR should be corrected at the time of Coronary artery bypass grafting(CABG).

Surgical correction of moderate IMR at the time of coronary revascularization is still an unresolved controversy.CABG alone did reduce MR at follow-up; nevertheless, CABG alone cannot be sufficient to eliminate MR in all cases , Adding mitral valve annuloplasty to CABG may eliminate MR immediately after surgery; however, recurrent MR did occur after CABG plus mitral valve annuloplasty, and no benefit for long-term survival was observed. There was also a tendency toward higher morbidity and mortality in CABG plus mitral valve procedure as compared with CABG alone in high-risk patients with moderate IMR. The latest American Association for Thoracic Surgery (AATS)guidelines suggested that for moderate IMR, mitral valve repair with an undersized complete rigid ring annuloplasty "may be considered" during CABG surgery, but not necessarily "preferred" over revascularization alone.Therefore ,the benefits of adding mitral valve procedure to CABG for treating moderate IMR have not been clearly established.

This study is aiming to determine the short term morbidity in patients undergoing CABG alone and comparing them with patients undergoing concomitant MV repair by assessment of morbidity and mortality in both groups postoperatively .

ELIGIBILITY:
Inclusion Criteria:

* All patient with multi-vessel coronary artery disease with moderate degree of ischemic mitral regurgitation .
* Patient undergone surgery using cardiopulmonary bypass.
* Patient done on elective basis

Exclusion Criteria:

* CABG done by off-pump technique.
* patients not candidates for complete revascularization.
* patients with other valvular affection other than mitral valve.
* Patients done on emergency basis.
* patient known to have Rheumatic valvular heart disease.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: study will be conducted on all patients diagnosed as ischemic heart disease with multi-vessel disease indicated for CABG with moderate degree of ischemic mitral regurgitation and meeting inclusion and exclusion criteria at duration between 2019 and 2021 at cardiothoracic surgery department in Assuit university hospital
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-03 (Estimated); Primary Completion 2023-11 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
To compare the outcome of mitral valve repair plus CABG vs CABG alone. | post operative ECHO assessment after 6 months.
  the aim is to determine whether there is significant difference postoperatively in patients undergoing mitral valve repair+CABG and those with CABG only regarding post operative degree of MR.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamad Z Roushdi, PhD, Principal Investigator — Mzidane
Locations (1):
- Assiut university Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] 1. Magne J, Senechal M, Dumesnil JD, Pibarot P. Ischemic mitral regurgitation: a complex multifaceted disease. Cardiology.2009;112:244-59. 2. Loperfido F, Biasucci LM, Pennestri F, Laurenzi F, Gimigliano F, Vigna C, et al. Pulsed Doppler echocardiographic analysis of mitral regurgitation after myocardial infarction. Am J Cardiol.1986;58:692-7. 3. Otsuji Y, Kumanohoso T, Yoshifuku S, Matsukida K, Koriyama C, Kisanuki A, et al. Isolated annular dilatation does not usually cause important functional mitral regurgitation: comparison between patients with lone atrial fibrillation and those with idiopathic or ischemic cardiomyopathy. J Am Coll Cardiol.2002;15(39):1651-6. 4.Levine RA, Schwammenthal E. Ischemic mitral regurgitation on the threshold of a solution: from paradoxes to unifying concepts. Circulation. 2005;112:745-58. 5.Lam BK, Gilinov AM, Blackstone EH, Rajeswaran J, Yuh B, et al. Importance of ischemic mitral regurgitation. Ann Thorac Surg.2005;79:462-70. 6.Bax JJ, Braun J, Somer ST, Klautz R, Holman ER, Versteegh MI, et al. Restrictive annuloplasty and coronary revascularization in ischemic mitral regurgitation results in reverse left ventricular remodeling. Circulation. 2004;110:103-8. 7.Sandoval Y, Sorajja P, Harris KM. Contemporary management of ischemic mitral regurgitation: a review. Am J Med 2018;131: 887-95. 8.Malhotra A, Ananthanarayanan C, Wadhawa V, et al. OPCABG for moderate CIMR in elderly patients: a superior option? Braz J Cardiovasc Surg 2018; 33: 15-22. 9.Salmasi MY, Harky A, Chowdhury MF, et al. Should the mitral valve be repaired for moderate ischemic mitral regurgitation at the time of revascularization surgery? J Card Surg 2018; 33:374-84. 10.Chan KM, Punjabi PP, Flather M, et al. Coronary artery bypass surgery with or without mitral valve annuloplasty in moderate functional ischemic mitral regurgitation: final results of the Randomized Ischemic Mitral Evaluation (RIME) trial. Circulation 2012; 126: 2502-10. 11.Sun X, Huang J, Shi M, Huang G, Pang L, Wang Y. Predictors of moderate ischemic mitral regurgitation improvement after off-pump coronary artery bypass. J Thorac Cardiovasc Surg 2015; 149: 1606-12. 12.Rabbah JP, Siefert AW, Bolling SF,Yoganathan AP. Mitral valve annuloplasty and anterior leaflet augmentation for functional ischemic mitral regurgitation: quantitative comparison of coaptation and subvalvular tethering. J Thorac Cardiovasc Surg 2014;148: 1688-93. 13.Smith PK, Puskas JD, Ascheim DD, et al. Surgical treatment of moderate ischemic mitral regurgitation. N Engl J Med 2014;371: 2178-88. 14.Kron IL, LaPar DJ, Acker MA, et al. 2016 update to TheAmerican Association for Thoracic Surgery consensus guidelines:Ischemic mitral valve regurgitation. J,Thorac Cardiovasc Surg 2017; 153: 1076-9.